CLINICAL TRIAL: NCT05940155
Title: Pattern of Admission of Children With COVID-19 Admitted in Assuit University Children Hospital.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Hussien, assistant lecturer, Assiut University
Other Study IDs: Diagnosis of COVID-19
Record Dates: First submitted 2023-07-09; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Assess the Outcome for Children With Covid-19 Admitted in Assuit University Children Hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- mild cases
- moderate cases
  Interventions: Diagnostic Test: RT PCR test of COVID 19
- severe cases
  Interventions: Diagnostic Test: RT PCR test of COVID 19

INTERVENTIONS:
Diagnostic Test: RT PCR test of COVID 19 — diagnostic test by naso-pharyngel swab to confirm the diagnosis of covid-19 at moderate and severe cases.
  Groups: moderate cases; severe cases

SUMMARY:
A novel coronavirus was identified following a cluster of cases of pneumonia in Wuhan, China, in December 2019. It rapidly spread as an outbreak there. On the 23rd of January 2020, it was announced that the outbreak constituted apublic health emergency of international concern. Few weeks later, virus spread was recorded worldwide and was announcedas a pandemic by WHO in March 11, 2020.Global spread included Egypt, and the first case was recorded inEgypt onFebruary 14, 2020.Diagnosis of COVID-19 depend on a case definition of suspected and confirmed case.

Implementation of case definition depend on the clinical presentation of the case and on laboratory test as well asradiological finding.The cases will be stratified according to these collective data to different grades of severity.

Mild cases are either asymptomatic or symptomatic with Leucopenia and/or lymphopenia with no radiological evidence of pneumonia (upper respiratory tract illness ± one of the following symptoms: fever < 38, cough,GIT symptoms, myalgia and/or arthralgia).

Moderate cases include patients with leucopenia and/or lymphopenia with clinical and radiological evidence of pneumonia, including fever > 38 °Cwith or without cough and tachypnea (respiratory rate > 60 breaths/min forinfants < 2 months, > 50 breaths/min for infants 2-12 months, > 40 breaths/min for children 1-4 years, > 30 breaths/min for children older than5 years old), and the condition may be associated by moderate to severe dehydration.

Cases are considered as severe and critically ill if any of the following is present: - O2 saturation ≤ 92% despite escalating O2 therapy to maximal allowed 6 L/min - O2 saturation ≤ 90 % at room air - If the patient in septic shock, confused or hemodynamically unstable despite fluid resuscitation - If respiratory manifestations are combined with other organ failure - Chest radiography > 50% lesion or progressive lesion within 24-48 hrs.

Children may play a major role in community-based viral transmission. Available data suggest that children may have more upper respiratory tract involvement (including nasopharyngeal carriage) rather than lower respiratory tract involvement.

The decision of the site of management either at home or in hospital depends on the clinical presentation, requirement for supportive care, potential risk factors for severe disease, and the ability of the patient to self-isolate at home. Supportive treatment including sufficient fluid and calories intake, and additional oxygen supplementation should be used in the treatment of children infected with COVID-19. The aim is to prevent ARDS, organ failure, and secondary nosocomial infections. If bacterial infection is suspected, broad-spectrum antibiotics may be used.

ELIGIBILITY:
Inclusion Criteria:

* All the patients from birth up to 18 years old admitted with suspectedor confirmed cases of covid-19 in AUCH.

Exclusion Criteria:

* : Any patient not suspected or confirmed to have COVID-19

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All subjects that meet the selection criteria (suspectedor confirmed cases of covid-19) in the period from 1st April 2022 till 31th March 2023, examined and/or admitted in AUCH.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluate pattern of admission of children with covid-19 admitted in Assuit University Children Hospital. | one year
  Evaluate pattern of admission of children with covid-19 admitted in Assuit University Children Hospital.

SECONDARY OUTCOMES:
- Assess the outcome for children with covid-19 admitted in Assuit University Children Hospital | one year
  - Assess the outcome for children with covid-19 admitted in Assuit University Children Hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine and Surgery At Assiut Univesity, Asyut, Egypt